CLINICAL TRIAL: NCT04007367
Title: A Phase 3, Randomized, Double-Blind, Placebo-controlled Study of the Efficacy and Safety of SAGE-217 With a Fixed, Repeated Treatment Regimen on Relapse Prevention in Adults With Major Depressive Disorder
Brief Title: A Study to Evaluate SAGE-217 for Prevention of Relapse in Adult Participants With Major Depressive Disorder
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Internal company decision
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 217-MDD-302; 2019-002640-25 (EudraCT Number)
Record Dates: First submitted 2019-07-02; First posted 2019-07-05 (Actual); Results first posted 2022-10-03 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Major Depressive Disorder
Keywords: MDD; SAGE-217
MeSH Terms: conditions — Depressive Disorder, Major | interventions — zuranolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Open-Label Phase: SAGE-217 (Experimental): Participants self-administered SAGE-217, 30 milligrams (mg), oral capsule, once daily (QD) in the evening from Day 1 to Day 14.
  Interventions: Drug: SAGE-217
- Double-Blind Phase: Placebo (Placebo Comparator): Following the OL Phase, participants who exhibited a Hamilton Rating Scale for Depression (HAM-D) response, defined as a greater than or equal to (≥) 50% reduction from baseline in HAM-D total score were to be randomized to receive SAGE-217 matching placebo capsule, orally, QD, in the evening, in a total of five, 14-day treatment periods, each separated by a 6-week follow-up period during the 40-week DB Phase of the study. However, no participants were randomized to receive SAGE-217 matching placebo due to early study termination.
  Interventions: Drug: Placebo
- Double-Blind Phase: SAGE-217 (Experimental): Following the OL Phase, participants who exhibited a HAM-D response defined as a ≥ 50% reduction from baseline in HAM-D total score to SAGE-217 were randomized to receive SAGE-217, 30 mg, oral capsule, QD, in the evening, up to study termination date (i.e., up to approximately 22 weeks) during the DB Phase of the study.
  Interventions: Drug: SAGE-217

INTERVENTIONS:
Drug: SAGE-217 — SAGE-217 capsule
  Arms: Double-Blind Phase: SAGE-217; Open-Label Phase: SAGE-217
Drug: Placebo — SAGE-217 matching placebo capsule
  Arms: Double-Blind Phase: Placebo

SUMMARY:
This is a study with an Open-Label (OL) phase followed by a randomized, Double-Blind (DB), placebo-controlled phase to assess efficacy and safety of SAGE-217 on relapse prevention in adults with major depressive disorder (MDD).

DETAILED DESCRIPTION:
This study was previously posted by Sage Therapeutics. In November 2023, sponsorship of the trial was transferred to Biogen.

ELIGIBILITY:
Inclusion Criteria:

1. Participant had a diagnosis of MDD as diagnosed by Structured Clinical Interview for Diagnostic and DSM-5 Clinical Trial Version (SCID-5-CT), with symptoms that had been present for at least a 4-week period.
2. Participant had at least 1 prior major depressive episode (MDE) in the 5 years prior to Screening (not including the current episode).
3. Participant was willing to delay the start of any antidepressant, anxiolytic, insomnia, psychostimulant, prescription opioid regimens, and new psychotherapy (including Cognitive Behavioral Therapy for Insomnia [CBT-I]) until after study completion.

Exclusion Criteria:

1. Participant had attempted suicide associated with the current episode of MDD.
2. Participant had treatment-resistant depression, defined as persistent depressive symptoms despite treatment with adequate doses of antidepressants within the current major depressive episode (excluding antipsychotics) from two different classes for at least 4 weeks of treatment. Massachusetts General Hospital Antidepressant Treatment Response Questionnaire (MGH ATRQ) was used for this purpose.
3. Participant had a positive pregnancy test at screening or on Day 1 prior to dosing.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2019-08-06 (Actual); Primary Completion 2020-01-06 (Actual); Study Completion 2020-01-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (43):
- United States (43):
  - Sage Investigational Site, Bentonville, Arkansas
  - Sage Investigational Site, Bellflower, California
  - Sage Investigational Site, Garden Grove, California
  - Sage Investigational Site, Lemon Grove, California
  - Sage Investigational Site, Oceanside, California
  - Sage Investigational Site, Orange, California
  - Sage Investigational Site, Riverside, California
  - Sage Investigational Site, San Diego, California
  - Sage Investigational Site, San Marcos, California
  - Sage Investigational Site, Sherman Oaks, California
  - Sage Investigational Site, Coral Springs, Florida
  - Sage Investigational Site, Jacksonville, Florida
  - Sage Investigational Site, Lauderhill, Florida
  - Sage Investigational Site, Orlando, Florida
  - Sage Investigational Site, Alpharetta, Georgia
  - Sage Investigational Site, Atlanta, Georgia
  - Sage Investigational Site, Decatur, Georgia
  - Sage Investigational Site, Chicago, Illinois
  - Sage Investigational Site, Lincolnwood, Illinois
  - Sage Investigational Site, Lake Charles, Louisiana
  - Sage Investigational Site, Gaithersburg, Maryland
  - Sage Investigational Site, Boston, Massachusetts
  - Sage Investigational Site, Methuen, Massachusetts
  - Sage Investigational Site, Watertown, Massachusetts
  - Sage Investigational Site, Ann Arbor, Michigan
  - Sage Investigational Site, Las Vegas, Nevada
  - Sage Investigational Site, Berlin, New Jersey
  - Sage Investigational Site, Cherry Hill, New Jersey
  - Sage Investigational Site, Marlton, New Jersey
  - Sage Investigational Site, Albuquerque, New Mexico
  - Sage Investigational Site, Jamaica, New York
  - Sage Investigational Site, New York, New York
  - Sage Investigational Site, Rochester, New York
  - Sage Investigational Site, Dayton, Ohio
  - Sage Investigational Site, North Canton, Ohio
  - Sage Investigational Site, Oklahoma City, Oklahoma
  - Sage Investigational Site, Allentown, Pennsylvania
  - Sage Investigational Site, Memphis, Tennessee
  - Sage Investigational Site, Austin, Texas
  - Sage Investigational Site, Dallas, Texas
  - Sage Investigational Site, Richardson, Texas
  - Sage Investigational Site, Wichita Falls, Texas
  - Sage Investigational Site, Everett, Washington

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in this study at 28 investigative sites in the United States from 06 August 2019 to 06 January 2020.
Pre-assignment Details: The study was conducted in 2 parts: Open-Label (OL) and Double-Blind (DB) Phase. Participants received SAGE-217 during treatment period in OL Phase. Participants who exhibited a Hamilton Rating Scale for Depression response in OL Phase were to be randomized in a ratio of 1:1 to receive either SAGE-217 matching placebo or SAGE-217 oral capsule in DB Phase. However, the study was terminated by sponsor due to business decisions and only 2 participants entered the DB Phase and did not complete it.
Groups:
- Double-Blind Phase: Placebo: Following the OL Phase, participants who exhibited a Hamilton Rating Scale for Depression (HAM-D) response defined as a greater than or equal to (≥) 50% reduction from baseline in HAM-D total score were to be randomized to receive SAGE-217 matching placebo capsule, orally, QD, in the evening, in a total of five, 14-day treatment periods, each separated by a 6-week follow-up period during the 40-week DB Phase of the study. However, no participants were randomized to receive SAGE-217 matching placebo due to early study termination.
- Double-Blind Phase: SAGE-217: Following the OL Phase, participants who exhibited a HAM-D response, defined as a ≥ 50% reduction from baseline in HAM-D total score to SAGE-217 were randomized to receive SAGE-217, 30 mg, oral capsule, QD, in the evening, up to study termination date (i.e., up to approximately 22 weeks) during the DB Phase of the study.
Period: Open-Label Phase (8-Weeks)
Arm/Group | Open-Label Phase: SAGE-217 | Double-Blind Phase: Placebo | Double-Blind Phase: SAGE-217
Started | 53 | 0 | 0
Completed | 5 | 0 | 0
Not Completed | 48 | 0 | 0
Not completed — Study Terminated by Sponsor | 43 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0
Not completed — Withdrawal by Participant | 2 | 0 | 0
Not completed — Non-compliance | 1 | 0 | 0
Period: Double-Blind Phase (14-Weeks)
Arm/Group | Open-Label Phase: SAGE-217 | Double-Blind Phase: Placebo | Double-Blind Phase: SAGE-217
Started (Of the five participants who completed the OL Phase, only those participants who meet the randomization criteria for the DB Phase entered it.) | 0 | 0 | 2
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 2
Not completed — Withdrawal by Participant | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Safety Set included all participants who were administered the study drug.
Groups:
- Open-Label Phase: SAGE-217: Participants self-administered SAGE-217, 30 mg, oral capsule, QD in the evening from Day 1 to Day 14.
Arm/Group | Open-Label Phase: SAGE-217
Number analyzed (Participants) | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.6 (12.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 45
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 37
  More than one race | 3
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Time to Relapse During the DB Phase
Description: Time to relapse was defined as days from the first dose of the study drug in the DB Phase to the day of relapse during the DB Phase. Participant was considered to have relapsed if: 2 consecutive HAM-D scores were ≥ 18 assessed 7 to 14 days apart, any worsening of depression requiring hospitalization, Investigator-determined risk of suicide, or any other clinically relevant event whether or not hospitalization was required. HAM-D is a scale used to rate depression in participants who were already diagnosed as depressed. The HAM-D total score comprised a sum of 17 individual item scores. Items scored in a range of 0 to 2 included: insomnia, somatic symptoms, genital symptoms, loss of weight, and insight. Items scored in a range of 0 to 4 included: agitation, depressed mood, feelings of guilt, suicide, work and activities, retardation, anxiety, hypochondriasis. The HAM-D total score could range from 0 (not depressed) to 52 (severely depressed). Higher scores indicated more depression.
Time Frame: Day 56 (Day 1 of DB Phase) up to Day 153 (i.e., up to 22 weeks)
Population: Due to early termination of the study by the sponsor, no data was collected, and no efficacy analysis was performed as planned, thus data is not available for this outcome measure.
Groups:
- Double-Blind Phase: Placebo: Following the OL Phase, participants who exhibited a HAM-D response defined as a ≥ 50% reduction from baseline in HAM-D total score were to be randomized to receive SAGE-217 matching placebo capsule, orally, QD, in the evening, in a total of five, 14-day treatment periods, each separated by a 6-week follow-up period during the 40-week DB Phase of the study. However, no participants were randomized to receive SAGE-217 matching placebo due to early study termination.
Arm/Group | Double-Blind Phase: Placebo | Double-Blind Phase: SAGE-217
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Percentage of Participants Who Relapsed During the DB Phase
Description: Participant was considered to have relapsed if: 2 consecutive HAM-D scores were ≥ 18 assessed 7 to 14 days apart, worsening of depression requiring hospitalization, Investigator-determined risk of suicide, or other clinically relevant events whether hospitalization was required. HAM-D scale was used to rate depression in participants who were diagnosed as depressed. Total score is a sum of 17 individual item scores. Items in a range of 0-2 included: insomnia (early, middle, late), somatic symptoms (gastrointestinal and general), genital symptoms, loss of weight, and insight. Items in a range of 0-4 included: agitation, depressed mood (sadness, hopeless, helpless, worthless), feelings of guilt, suicide, work and activities, retardation (slowness of thought and speech; impaired ability to concentrate; decreased motor activity), anxiety (psychic and somatic), hypochondriasis. Total score could range from 0 (not depressed)- 52 (severely depressed). Higher scores indicated more depression.
Time Frame: Day 56 (Day 1 of DB Phase) up to Day 153 (i.e., up to 22 weeks)
Population: as for outcome 1
Arm/Group | Double-Blind Phase: Placebo | Double-Blind Phase: SAGE-217
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change From Baseline in the 17-Item HAM-D Total Score at the End of Each 14-Day Treatment Period in the DB Phase
Description: The 17-item HAM-D scale was used to rate the severity of depression in participants who were already diagnosed as depressed. The HAM-D total score comprised a sum of 17 individual item scores. Items scored in a range of 0 to 2 included: insomnia (early, middle, late), somatic symptoms (gastrointestinal and general), genital symptoms, loss of weight, and insight. Items scored in a range of 0 to 4 included: agitation, depressed mood (sadness, hopeless, helpless, worthless), feelings of guilt, suicide, work and activities, retardation (slowness of thought and speech; impaired ability to concentrate; decreased motor activity), anxiety (psychic and somatic), hypochondriasis. The HAM-D total score could range from 0 (not depressed) to 52 (severely depressed). Higher scores indicated more depression. A negative change from baseline indicated improvement.
Time Frame: Day 56 (Baseline [Day 1] of DB Phase) up to Day 153 (i.e., up to 22 weeks)
Population: as for outcome 1
Arm/Group | Double-Blind Phase: Placebo | Double-Blind Phase: SAGE-217
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Percentage of Participants With HAM-D Response at the End of Each 14-Day Treatment Period in the DB Phase
Description: HAM-D response was defined as having a 50% or greater reduction from baseline in HAM-D total score. The HAM-D total score comprised a sum of 17 individual item scores. Items scored in a range of 0 to 2 included: insomnia (early, middle, late), somatic symptoms (gastrointestinal and general), genital symptoms, loss of weight, and insight. Items scored in a range of 0 to 4 included: agitation, depressed mood (sadness, hopeless, helpless, worthless), feelings of guilt, suicide, work and activities, retardation (slowness of thought and speech; impaired ability to concentrate; decreased motor activity), anxiety (psychic and somatic), hypochondriasis. The HAM-D total score could range from 0 (not depressed) to 52 (severely depressed). Higher scores indicated more depression.
Time Frame: Day 56 (Day 1 of DB Phase) up to Day 153 (i.e., up to 22 weeks)
Population: as for outcome 1
Arm/Group | Double-Blind Phase: Placebo | Double-Blind Phase: SAGE-217
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Percentage of Participants With HAM-D Remission at the End of Each 14-Day Treatment Period in the DB Phase
Description: HAM-D remission was defined as having a HAM-D total score of ≤ 7. The HAM-D total score comprised a sum of 17 individual item scores. Items scored in a range of 0 to 2 included: insomnia (early, middle, late), somatic symptoms (gastrointestinal and general), genital symptoms, loss of weight, and insight. Items scored in a range of 0 to 4 included: agitation, depressed mood (sadness, hopeless, helpless, worthless), feelings of guilt, suicide, work and activities, retardation (slowness of thought and speech; impaired ability to concentrate; decreased motor activity), anxiety (psychic and somatic), hypochondriasis. The HAM-D total score could range from 0 (not depressed) to 52 (severely depressed). Higher scores indicated more depression.
Time Frame: Day 56 (Day 1 of DB Phase) up to Day 153 (i.e., up to 22 weeks)
Population: as for outcome 1
Arm/Group | Double-Blind Phase: Placebo | Double-Blind Phase: SAGE-217
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Percentage of Participants With Clinical Global Impression - Improvement (CGI-I) Response at the End of Each 14-Day Treatment Period in the DB Phase
Description: The CGI-I employs a 7-point Likert scale to measure the overall improvement in the participant's condition posttreatment. The Investigator rated the participant's total improvement whether or not it was due entirely to drug treatment. Response choices included: 1=very much improved, 2=much improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=much worse, and 7=very much worse. The CGI-I is only rated at posttreatment assessments. By definition, all CGI-I assessments are evaluated against baseline conditions. Higher score indicated worse condition. CGI-I response was defined as having a CGI-I score of "very much improved" or "much improved."
Time Frame: Day 56 (Day 1 of DB Phase) up to Day 153 (i.e., up to 22 weeks)
Population: as for outcome 1
Arm/Group | Double-Blind Phase: Placebo | Double-Blind Phase: SAGE-217
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change From Baseline in Clinical Global Impression - Severity (CGI-S) Score at the End of Each 14-Day Treatment Period in the DB Phase
Description: The CGI-S uses a 7-point Likert scale to rate the severity of the participant's illness at the time of assessment, relative to the clinician's past experience with participants who had the same diagnosis. Considering total clinical experience, a participant was assessed on severity of mental illness at the time of rating as 1=normal, not at all ill; 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; and 7= among the most extremely ill participant. A higher score indicated extreme illness. A negative change from baseline indicated improvement (a higher absolute number indicating more illness).
Time Frame: Day 56 (Baseline [Day 1] of DB Phase) up to Day 153 (i.e., up to 22 weeks)
Population: as for outcome 1
Arm/Group | Double-Blind Phase: Placebo | Double-Blind Phase: SAGE-217
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change From Baseline in 9-Item Patient Health Questionnaire (PHQ-9) Score at the End of Each 14-Day Treatment Period in the DB Phase
Description: The PHQ-9 is a participant-rated depressive symptom severity scale. To monitor severity over time participants in current treatment for depression, participants completed the questionnaires at baseline and at regular intervals thereafter. Scoring was based on responses to specific questions, as follows: 0=not at all; 1=several days; 2=more than half the days; and 3=nearly every day. The PHQ-9 total score was calculated as the sum of the 9 individual item scores and ranged from 0 to 27. The PHQ-9 total score was categorized as follows: 1 to 4=minimal depression, 5 to 9=mild depression, 10 to 14=moderate depression, 15 to 19=moderately severe depression; and 20 to 27=severe depression. Higher score indicated severe depression. A negative change from baseline indicated improvement.
Time Frame: Day 56 (Baseline [Day 1] of DB Phase) up to Day 153 (i.e, up to 22 weeks)
Population: as for outcome 1
Arm/Group | Double-Blind Phase: Placebo | Double-Blind Phase: SAGE-217
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Time to Relapse During The DB Phase for Participants Who Achieved HAM-D Remission in the OL Phase
Description: Time to relapse was defined as days from the first dose of the study drug in the DB Phase to the day of relapse during the DB Phase. Participant was considered to have relapsed if: 2 consecutive HAM-D scores were ≥18 assessed 7 to 14 days apart, any worsening of depression requiring hospitalization, Investigator-determined risk of suicide, or any other clinically relevant event whether or not hospitalization was required. HAM-D is a scale used to rate depression in participants who were already diagnosed as depressed. The HAM-D total score comprised a sum of 17 individual item scores. Items scored in a range of 0 to 2 included: insomnia, somatic symptoms, genital symptoms, loss of weight, and insight. Items scored in a range of 0 to 4 included: agitation, depressed mood, feelings of guilt, suicide, work and activities, retardation, anxiety, hypochondriasis. The HAM-D total score could range from 0 (not depressed) to 52 (severely depressed). Higher scores indicated more depression.
Time Frame: Day 56 (Day 1 of DB Phase) up to Day 153 (i.e., up to 22 weeks)
Population: as for outcome 1
Arm/Group | Double-Blind Phase: Placebo | Double-Blind Phase: SAGE-217
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. A TEAE was defined as an AE with onset after the start of study drug, or any worsening of a pre-existing medical condition/AE with onset after the start of study drug and throughout the study.
Time Frame: From the first dose of study drug up to the end of the study (i.e., up to approximately 22 weeks)
Population: Safety Set included all participants who were administered the study drug. Data for this outcome measure was not collected for DB Phase: Placebo arm because none of the participants were enrolled into this group.
Measure: Count of Participants; unit: Participants
Groups:
- Double-Blind Phase: Placebo: Following the OL Phase participants who exhibited a HAM-D response defined as a ≥ 50% reduction from baseline in HAM-D total score were to be randomized to receive SAGE-217 matching placebo capsule, orally, QD, in the evening, in a total of five, 14-day treatment periods, each separated by a 6-week follow-up period during the 40-week DB Phase of the study. However, no participants were randomized to receive SAGE-217 matching placebo due to early study termination.
Arm/Group | Open-Label Phase: SAGE-217 | Double-Blind Phase: Placebo | Double-Blind Phase: SAGE-217
Number analyzed (Participants) | 53 | 0 | 2
Participants | 26 |  | 0

ADVERSE EVENTS:
Time Frame: From the first dose of study drug up to the end of the study (i.e., up to approximately 22 weeks)
Description: Safety Set included all participants who were administered the study drug. Safety data for the placebo arm in the DB phase was not collected because none of the participants were enrolled in this group.
Arm/Group | Open-Label Phase: SAGE-217 | Double-Blind Phase: Placebo | Double-Blind Phase: SAGE-217
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/0 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/0 | 0/2
Other Adverse Events (participants affected / at risk) | 19/53 | 0/0 | 0/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Open-Label Phase: SAGE-217 (N=53) | Double-Blind Phase: Placebo (N=0) | Double-Blind Phase: SAGE-217 (N=2)
Vomiting (Gastrointestinal disorders) | 3 | 0 | 0
Dizziness (Nervous system disorders) | 3 | 0 | 0
Headache (Nervous system disorders) | 5 | 0 | 0
Sedation (Nervous system disorders) | 4 | 0 | 0
Somnolence (Nervous system disorders) | 4 | 0 | 0

LIMITATIONS AND CAVEATS:
The study was stopped prematurely and therefore data was not collected and analyzed for any efficacy outcome measure planned for the DB Phase of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for non-commercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2019-08-29): https://cdn.clinicaltrials.gov/large-docs/67/NCT04007367/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-23): https://cdn.clinicaltrials.gov/large-docs/67/NCT04007367/SAP_001.pdf